CLINICAL TRIAL: NCT03301987
Title: Therapeutic Exercise in Patients With Chronic Kidney Disease
Brief Title: Chronic Kidney Disease & Therapeutic Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de León (Other)
Responsible Party: Principal Investigator, César Calvo Lobo, PhD, MSc, PT, Universidad de León
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERC_ULE
Record Dates: First submitted 2017-09-30; First posted 2017-10-04 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Kidney; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeutic exercise (Experimental)
  Interventions: Other: Therapeutic exercise

INTERVENTIONS:
Other: Therapeutic exercise — 30 minutes per day of therapeutic exercise

SUMMARY:
The aim of this study is to evaluate the therapeutic exercise effects in patients with chronic kidney disease. An interventional prospective study is carried out. A sample of 9 patients with chronic kidney disease is recruited. The kidney function (creatinine clearance as main outcome) is measured at baseline and 1 month after treatment start.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic kidney disease

Exclusion Criteria:

* Cognitive impairment and non signed consent inform form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-10-14 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2017-12-09 (Actual)

PRIMARY OUTCOMES:
Kidney function | Change from Baseline creatinine clearance at 1 month
  Creatinine clearance

CONTACTS AND LOCATIONS:
Locations (1):
- Pierre Neyra Bohórquez, Galdakao, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Calvo-Lobo C, Neyra-Bohorquez PP, Seco-Calvo J. Aerobic exercise effects in renal function and quality of life of patients with advanced chronic kidney disease. Rev Assoc Med Bras (1992). 2019 Jun 3;65(5):657-662. doi: 10.1590/1806-9282.65.5.657. PMID 31166442